CLINICAL TRIAL: NCT04831814
Title: Near-focus Versus Normal-focus Narrow Band Imaging Colonoscopy in Diagnosis of Colorectal Polyps Based on Combined NICE and WASP Classification: a Randomized Controlled Trial
Brief Title: Narrow Band Imaging in Diagnosis of Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, Principal Investigation, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 61355143
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Polyp; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near Focus NBI (Experimental): Use of the Near Focus NBI to make optical diagnosis
  Interventions: Diagnostic Test: Near Focus NBI
- Standard Focus NBI (Active Comparator): Use of the Standard Focus NBI to make optical diagnosis
  Interventions: Diagnostic Test: Standard Focus NBI

INTERVENTIONS:
Diagnostic Test: Near Focus NBI — Colonoscopy with near focus narrowing band imaging technology . Optical specifications include a 2 mm near field focal depth. Optical diagnosis of polyps were according to NICE and WASP, respectively.
  Arms: Near Focus NBI
Diagnostic Test: Standard Focus NBI — Colonoscopy with narrow band imaging technology.Optical diagnosis of polyps were according to NICE and WASP, respectively.
  Arms: Standard Focus NBI

SUMMARY:
Optical diagnosis of colorectal polyps is a promising tool to avoid risks of unnecessary polypectomies and to save costs of tissue pathology. NICE (NBI International Colorectal Endoscopic) and WASP (Workgroup on Serrated Polyps and Polyposis) classification were developed for diagnosis of adenomatous and sessile serrated polyps, respectively.

DETAILED DESCRIPTION:
Near-focus (NF) narrow-band imaging (NBI) is an image-magnifying technology which enables optical magnification of up to 65x in near focus (NF) compared with 52x in normal standard focus (SF) with the simple push of a button of the endoscope to be interchangeable between NF and SF. There were few studies comparing diagnostic accuracy between NF and SF in the diagnosis of colorectal polyps. So, our aim of the current study is to compare accuracy of NF NBI compared with SF NBI in the optical diagnosis of neoplastic and non-neoplastic polyp and the accuracy of NF NBI versus SF NBI in distinguishing serrated adenoma from hyperplastic polyp in sessile lesions using histologic evaluation as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for colonoscopy at NKC institute

Exclusion Criteria:

* Inflammatory bowel disease
* Polyposis syndrome
* Colorectal cancer
* Active gastrointestinal bleeding
* Pregnant woman
* Inadequate bowel preparation
* Contraindication for polyps removal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Rate of accurate polyp histology predictions by the Endoscopists in the two groups. | At the time of procedure
  Measure of the percentage of accurate predictions by the endoscopists in the differentiation of neoplastic from non neoplastic colorectal lesions, using the high definition NBI colonoscopy with and without near focus features
Rate of accurate diagnosis of sessile serrated polyps/adenoma by the Endoscopists in the two groups. | At the time of procedure
  Measure of the percentage od accurate predictions by the endoscopists in the differentiation of sessile serrated polyps/adenoma from hyperplastic polyps, using the high definition NBI colonoscopy with and without near focus features.

SECONDARY OUTCOMES:
The polyp detection rate | At the time of procedure
  The prevalence of patients with at least one polyp was detected
The adenoma detection rate | At the time of procedure
  The prevalence of patients with at least one adenoma was detected
Diagnostic Characteristics | At the time of procedure
  Compare the diagnostic characteristic (sensitivity, specificity, positive predictive value and negative predictive value) using the high definition narrow band imaging colonoscopy with and without near focus features.

CONTACTS AND LOCATIONS:
Overall Officials: NISA NETINATSUNTON, MD., Principal Investigator — NKC Institute of Gastroenterology and Hepatology, Prince of Songkla University
Locations (1):
- Prince Songkla University, Hat Yai, Changwat Songkhla, Thailand